CLINICAL TRIAL: NCT03104491
Title: Inotuzumab Ozogamicin Post-Transplant For Acute Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leland Metheny (Other)
Responsible Party: Sponsor-Investigator, Leland Metheny, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1916
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: allogeneic hematopoietic stem cell transplantation; donor chimerism
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inotuzumab Ozogamicin (Experimental): Phase I:
  A maximum of 4 cycles will be allowed and doses will be adjusted in 0.1mg/m2 increments using a dose escalation scale depending on tolerability. Total range of dose levels for participants is 0.1-0.6mg/m^2.
  Phase II:
  Participants will be enrolled until all Phase I participants have been followed and assessed for toxicity for at least 4 weeks after the fourth treatment dose of inotuzumab ozogamicin or 4 weeks after the participant goes off treatment, whichever comes first. Doses to be administered will be determined in the phase I portion of the study. The recommended phase 2 dose is 0.3mg/m2. Repeat cycles every 28 days for up to 4 cycles
  Interventions: Drug: Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin — Inotuzumab ozogamicin, IV, 28 day cycles
  Phase 1 dosages:
  Dose Level -2 (0.1 mg/m^2)
  Dose Level -1 (0.2 mg/m^2)
  Dose Level 0 (0.3 mg/m^2)
  Dose Level 1 (0.4 mg/m^2)
  Dose Level 2 (0.5 mg/m^2)
  Dose Level 3 (0.6 mg/m^2)

SUMMARY:
This study has two phases, Phase I and Phase II. The main goal of the Phase I portion of this research study is to see what doses post-transplant inotuzumab ozogamicin can safely be given to subjects without having too many side effects.

The Phase II portion of this study is to see what side effects are seen with medication after transplant.

Inotuzumab ozogamicin is a combination of an antibody and chemotherapy which has been shown to have significant activity against relapsed/refractory acute lymphocytic leukemia (ALL).

Inotuzumab ozogamicin is considered experimental in this study.

DETAILED DESCRIPTION:
Study Design This is a Phase I/II study of inotuzumab ozogamicin for the treatment of patients who underwent allogeneic transplantation for ALL and have a high risk of relapse. The Phase I portion of this study will be a 3+3 dose escalation trial. This is followed by a phase 2 cohort at the recommended Phase 2 dose (RP2D). Participants will receive study treatment up to 4 cycles until relapse of disease, unacceptable toxicity, or death, whichever occurs first

Phase I: Inotuzumab Ozogamicin Dosing Escalation Subjects will be assessed for safety and tolerability (including adverse events, serious adverse events, and clinical/laboratory assessments) using a continuous monitoring approach.

Phase II: Inotuzumab Ozogamicin Subjects will be assessed for safety and tolerability (including adverse events, serious adverse events, and clinical/laboratory assessments) using a continuous monitoring approach. In order to be included in the safety profile endpoint review, subjects must have received at least of 1 cycle of treatment.

Primary Objective

Phase I: To define a post hematopoietic stem cell transplantation maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of inotuzumab ozogamicin.

Phase II: To assess the efficacy of inotuzumab ozogamicin as measured by diseasefree survival (DFS) at one year.

Secondary Objective(s)

Phase I:

* To evaluate disease-free survival (DFS), nonrelapse mortality (NRM), relapse, relapse-related mortality and overall survival (OS) at 1 year.
* To determine safety profile of inotuzumab ozogamicin after transplant including the incidence of myeloid toxicity and secondary graft failure and the rate of veno-occlusive disease/sinusoidal obstruction syndrome (VOD/SOS).
* To determine if inotuzumab ozogamicin at these doses is effective at eradicating minimal residual disease in this cohort of participants

Phase II:

* To assess additional evidence of efficacy and safety as measured by non-relapse mortality (NRM), relapse, relapse-related mortality and overall survival (OS) at 1 year.
* To determine if inotuzumab ozogamicin at these doses is effective at eradicating MRD.
* To confirm the safety profile of inotuzumab ozogamicin therapy after transplant including myeloid toxicity, secondary graft failure, and the rate of VOD/SOS.
* To evaluate the pharmacokinetics of inotuzumab ozogamicin post allogeneic transplant

ELIGIBILITY:
Inclusion Criteria:

Phase 1 Inclusion Criteria

* Diagnosis of CD22-positive Acute Lymphoblastic Leukemia
* Patients who underwent an allogeneic hematopoietic stem cell transplantation from any donor source for acute lymphocytic leukemia
* Patients who are between T+40 and T+100 after allogeneic transplantation. Patients must receive their first dose of inotuzumab at or before T+100.
* Patients who have/are either:

  * Transplanted in hematologic first complete remission with evidence of minimal residual disease within 45 days of allogeneic transplantation

    ---Pre- or Post-Transplant Minimal Residual Disease defined by:

    ----Any detectable ALL (by flow cytometry, cytogenetics, or PCR techniques) as per clinical indication.
  * In second or third complete remission at the time of allogeneic transplantation
  * Treated with reduced intensity regimens or non-myeloablative conditioning regimens
  * Lymphoid blast crisis of CML
  * Are relapsed or refractory to at least 1 line of chemotherapy
  * Philadelphia-like ALL
* Patients who have evidence of donor chimerism after allogeneic transplantation.
* ECOG Performance status < 2
* Participants must have ANC > 1,000/µL for 3 days and platelet transfusion independence as defined as a platelet count > 50,000/µL for 7 days.
* Able to adhere to the study visit schedule and other protocol requirements.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.

Phase 2 Inclusion Criteria

* Diagnosis of CD22-positive Acute Lymphoblastic Leukemia
* Patients who underwent an allogeneic hematopoietic stem cell transplantation from any donor source for acute lymphocytic leukemia
* Patients who are between T+40 and T+100 after allogeneic transplantation
* Patients who have/are either:

  * Transplanted in hematologic first complete remission with evidence of minimal residual disease within 45 days of allogeneic transplantation

    ---Post-Transplant Minimal Residual Disease defined by:

    ----Any detectable ALL (by flow cytometry, cytogenetics, or PCR techniques) as per clinical indication.
  * In second or third complete remission at the time of allogeneic transplantation
  * Treated with reduced intensity regimens as defined per institutional standard of practice
  * Lymphoid blast crisis of CML
  * Are relapsed or refractory to at least 1 line of chemotherapy
  * Philadelphia-like ALL
* Patients who have > 80% donor chimerism after allogeneic transplantation.
* Philadelphia chromosome positive ALL must have failed at least 1 TKI
* ECOG Performance status < 1
* pre-transplant evaluation, see 10.1.1
* Participants must have ANC > 1,000/µL for 3 days and platelet transfusion independence as defined as a platelet count > 50,000/µL for 7 days.
* Able to adhere to the study visit schedule and other protocol requirements.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.

Phase 1 and 2 Exclusion Criteria:

* Patients with clinical evidence of disease progression prior to enrollment
* Persistent prior treatment toxicities Grade 2 and above according to NCI CTCAE Version 4.03 (with the exception for alopecia, neuropathy, etc.)
* Patients with inadequate organ function as defined by:

  * Creatinine clearance < 30ml/min
  * Bilirubin > 2X institutional upper limit of normal
  * AST (SGOT) > 2X institutional upper limit of normal
  * ALT (SGPT) > 2X institutional upper limit of normal
* GVHD grade III or IV (for patients with a prior allogeneic transplant).
* Active acute or chronic GVHD of the liver (for patients with a prior allogeneic transplant)
* History of VOD
* Use of concomitant TKI or sirolimus
* Second active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast)
* Patients with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because inotuzumab ozogamicin may be associated with the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with inotuzumab ozogamicin, breastfeeding should be discontinued if the mother is treated with inotuzumab ozogamicin. These potential risks may also apply to other agents used in this study.
* Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.)
* Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.)
* Participation in any other investigational drug study or had exposure to any other investigational agent, device, or procedure, within 21 days (or 5 half-lives, whichever is greater)
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Phase I MTD | Up to 112 days (16 weeks)
  Defined post hematopoietic stem cell transplantation MTD
Phase I DLTs | Up to 112 days (16 weeks)
  Frequency of DLTs during the first two cycles in ALL-participants
Phase II Median DFS | At 3 months after initial treatment
  Efficacy as measured by phase II DFS at one year, estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)".
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
  In Phase II, the null hypothesis of H0: DFS at 1-year ≤ 55% versus the alternative hypothesis of Ha: DFS at 1-year ≥ 75% using 1-sided alpha of 10% will be tested
Phase II Median DFS | At 6 months after initial treatment
  Efficacy as measured by phase II DFS at one year, estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)".
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
  In Phase II, the null hypothesis of H0: DFS at 1-year ≤ 55% versus the alternative hypothesis of Ha: DFS at 1-year ≥ 75% using 1-sided alpha of 10% will be tested
Phase II Median DFS | At 9 months after initial treatment
  Efficacy as measured by phase II DFS at one year, estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)".
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
  In Phase II, the null hypothesis of H0: DFS at 1-year ≤ 55% versus the alternative hypothesis of Ha: DFS at 1-year ≥ 75% using 1-sided alpha of 10% will be tested
Phase II Median DFS | At 1 year after initial treatment
  Efficacy as measured by phase II DFS at one year, estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)".
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
  In Phase II, the null hypothesis of H0: DFS at 1-year ≤ 55% versus the alternative hypothesis of Ha: DFS at 1-year ≥ 75% using 1-sided alpha of 10% will be tested
Phase II Median DFS | Post first dose of inotuzumab ozogamicin
  Efficacy as measured by phase II DFS at one year, estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)".
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
  In Phase II, the null hypothesis of H0: DFS at 1-year ≤ 55% versus the alternative hypothesis of Ha: DFS at 1-year ≥ 75% using 1-sided alpha of 10% will be tested

SECONDARY OUTCOMES:
Phase I Median DFS | At 3 months after initial treatment
  Efficacy as measured by phase I DFS at one year. Estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)"
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I Median DFS | At 6 months after initial treatment
  Efficacy as measured by phase I DFS at one year. Estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)"
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I Median DFS | At 9 months after initial treatment
  Efficacy as measured by phase I DFS at one year. Estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)"
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I Median DFS | At 1 year after initial treatment
  Efficacy as measured by phase I DFS at one year. Estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)"
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I Median DFS | Post first dose of inotuzumab ozogamicin on Day 1, Cycle 1, where cycle length is 28 days
  Efficacy as measured by phase I DFS at one year. Estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI)
  DFS is defined as "Time from date of first dose to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)"
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I NRM | At 3 months after initial treatment
  Phase I NRM, defined as time from date of first dose to death due to any cause without prior relapse. Criteria used: For ALL, evidence of disease in the blood or bone marrow (flow cytometry or PCR).
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I NRM | At 6 months after initial treatment
  Phase I NRM, defined as time from date of first dose to death due to any cause without prior relapse. Criteria used: For ALL, evidence of disease in the blood or bone marrow (flow cytometry or PCR).
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I NRM | At 9 months after initial treatment
  Phase I NRM, defined as time from date of first dose to death due to any cause without prior relapse. Criteria used: For ALL, evidence of disease in the blood or bone marrow (flow cytometry or PCR).
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I NRM | At 1 year after initial treatment
  Phase I NRM, defined as time from date of first dose to death due to any cause without prior relapse. Criteria used: For ALL, evidence of disease in the blood or bone marrow (flow cytometry or PCR).
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I NRM | Post first dose of inotuzumab ozogamicin on Day 1, Cycle 1, where cycle length is 28 days
  Phase I NRM , defined as time from date of first dose to death due to any cause without prior relapse. Criteria used: For ALL, evidence of disease in the blood or bone marrow (flow cytometry or PCR).
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse | At 3 months after initial treatment
  Phase I relapse rate, defined as time from date of first dose to the date of first relapse.
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse | At 6 months after initial treatment
  Phase I relapse rate, defined as time from date of first dose to the date of first relapse.
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse | At 9 months after initial treatment
  Phase I relapse rate, defined as time from date of first dose to the date of first relapse.
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse | At 1 year after initial treatment
  Phase I relapse rate, defined as time from date of first dose to the date of first relapse.
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse | Post first dose of inotuzumab ozogamicin on Day 1, Cycle 1, where cycle length is 28 days
  Phase I relapse rate, defined as time from date of first dose to the date of first relapse.
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse-related mortality | At 3 months after initial treatment
  Phase I Relapse-related mortality, defined time from date of first dose to death due to any cause with prior relapse
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse-related mortality | At 6 months after initial treatment
  Phase I Relapse-related mortality, defined time from date of first dose to death due to any cause with prior relapse
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse-related mortality | At 9 months after initial treatment
  Phase I Relapse-related mortality, defined time from date of first dose to death due to any cause with prior relapse
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse-related mortality | At 1 year after initial treatment
  Phase I Relapse-related mortality, defined time from date of first dose to death due to any cause with prior relapse
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Relapse-related mortality | Post first dose of inotuzumab ozogamicin on Day 1, Cycle 1, where cycle length is 28 days
  Phase I Relapse-related mortality, defined time from date of first dose to death due to any cause with prior relapse
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase I Median OS | At 3 months after initial treatment
  Phase I OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I Median OS | At 6 months after initial treatment
  Phase I OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I Median OS | At 9 months after initial treatment
  Phase I OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I Median OS | At 1 year after initial treatment
  Phase I OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I Median OS | Post first dose of inotuzumab ozogamicin on Day 1, Cycle 1, where cycle length is 28 days
  Phase I OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase I Incidence of myeloid toxicity | At 1 year
  Number of patients who develop myeloid toxicity while on study, defined as grade of anemia, neutropenia and thrombocytopenia CTCAE 4
Phase I Incidence of secondary graft failure | At 1 year
  Number of patients who develop secondary graft failure while on study, defined as:
  Either cytopenias after initial engraftment (ANC <500/µL), with (a) donor chimerism of less than 5% or (b) falling donor chimerism with intervention such as second transplant or donor lymphocyte infusion (DLI) or (c) patient death due to cytopenias, and fall in donor chimerism, even if chimerism was >5%. Exclusion criteria for diagnosis of GF were (a) disease relapse (b) graft versus host disease or (c) other causes of cytopenias such as, viral infections, or drug induced
Phase I incidence of veno-occlusive disease/sinusoidal obstruction syndrome (VOD/SOS) | At 1 year
  Safety profile of intervention as measured by incidence of VOD/SOS disease in the phase I portion of the study, defined as the occurrence of 2 of the following 3 clinical criteria:
  * Total serum bilirubin level >34 μmol/L (>2.0 mg/dL).
  * An increase in liver size from baseline or development of right upper quadrant pain of liver origin.
  * Sudden weight gain >2.5% during any 72-hour period after infusion of investigational product because of fluid accumulation or development of ascites.
Phase I rate of VOD/SOS - number of participants affected | At 1 year
  Safety profile of intervention as measured by number of participants affected by VOD/SOS disease in the phase I portion of the study, defined as the occurrence of 2 of the following 3 clinical criteria:
  * Total serum bilirubin level >34 μmol/L (>2.0 mg/dL).
  * An increase in liver size from baseline or development of right upper quadrant pain of liver origin.
  * Sudden weight gain >2.5% during any 72-hour period after infusion of investigational product because of fluid accumulation or development of ascites.
Phase I - Percent of participants with grade 3 + AE/SAEs | At 1 year
  Phase I safety profile of intervention as measured by percent of participants with grade 3 + AE/SAEs
Phase II Non-relapse mortality (NRM) | At 3 months after initial treatment
  Phase II Non-relapse mortality (NRM), defined as time from date of first dose to death due to any cause without prior relapse.
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase II Relapse | At 6 months after initial treatment
  Phase II relapse rate, defined as time from date of first dose to the date of first relapse.
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase II Relapse | At 9 months after initial treatment
  Phase II relapse rate, defined as time from date of first dose to the date of first relapse.
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase II Relapse-related mortality | At 1 year after initial treatment
  Phase II Relapse-related mortality, defined time from date of first dose to death due to any cause with prior relapse
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase II Relapse-related mortality | Post first dose of inotuzumab ozogamicin on Day 1, Cycle 1, where cycle length is 28 days
  Phase II Relapse-related mortality, defined time from date of first dose to death due to any cause with prior relapse
  Reported as Cumulative Incidence and 2-sided 80% CI and 2-sided 95% CI
Phase II Median OS | At 3 months after initial treatment
  Phase II OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase II Median OS | At 6 months after initial treatment
  Phase II OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase II Median OS | At 9 months after initial treatment
  Phase II OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase II Median OS | At 1 year after initial treatment
  Phase II OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase II Median OS | Post first dose of inotuzumab ozogamicin on Day 1, Cycle 1, where cycle length is 28 days
  Phase II OS, defined from time from date of first dose to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI
  Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Phase II Response Rate | At 3 months after initial treatment
  Defined as the proportion of patients with a best overall response of eradicating MRD at the time each patient discontinues treatment with Inotuzumab Ozogamicin
Phase II Response Rate | At 6 months after initial treatment
  Defined as the proportion of patients with a best overall response of eradicating MRD at the time each patient discontinues treatment with Inotuzumab Ozogamicin
Phase II Response Rate | At 9 months after initial treatment
  Defined as the proportion of patients with a best overall response of eradicating MRD at the time each patient discontinues treatment with Inotuzumab Ozogamicin
Phase II Response Rate | At 1 year after initial treatment
  Defined as the proportion of patients with a best overall response of eradicating MRD at the time each patient discontinues treatment with Inotuzumab Ozogamicin
Phase II Response Rate | Post first dose of inotuzumab ozogamicin on Day 1, Cycle 1, where cycle length is 28 days
  Defined as the proportion of patients with a best overall response of eradicating MRD at the time each patient discontinues treatment with Inotuzumab Ozogamicin
Phase II Incidence of myeloid toxicity | At 1 year
  Number of patients who develop myeloid toxicity while on study, defined as grade of anemia, neutropenia and thrombocytopenia CTCAE 4
Phase II Incidence of secondary graft failure | At 1 year after initial treatment
  Number of patients who develop secondary graft failure while on study, defined as:
  Either cytopenias after initial engraftment (ANC <500/µL), with (a) donor chimerism of less than 5% or (b) falling donor chimerism with intervention such as second transplant or donor lymphocyte infusion (DLI) or (c) patient death due to cytopenias, and fall in donor chimerism, even if chimerism was >5%. Exclusion criteria for diagnosis of GF were (a) disease relapse (b) graft versus host disease or (c) other causes of cytopenias such as, viral infections, or drug induced
Phase I incidence of VOD/SOS | At 1 year
  Safety profile of intervention as measured by incidence of VOD/SOS disease in the phase I portion of the study, defined as the occurrence of 2 of the following 3 clinical criteria:
  * Total serum bilirubin level >34 μmol/L (>2.0 mg/dL).
  * An increase in liver size from baseline or development of right upper quadrant pain of liver origin.
  * Sudden weight gain >2.5% during any 72-hour period after infusion of investigational product because of fluid accumulation or development of ascites.
Phase II rate of VOD/SOS - number of participants affected | At 1 year
  Safety profile of intervention as measured by number of participants affected by VOD/SOS disease in the phase I portion of the study, defined as the occurrence of 2 of the following 3 clinical criteria:
  * Total serum bilirubin level >34 μmol/L (>2.0 mg/dL).
  * An increase in liver size from baseline or development of right upper quadrant pain of liver origin.
  * Sudden weight gain >2.5% during any 72-hour period after infusion of investigational product because of fluid accumulation or development of ascites.
Phase II pharmacokinetic (PK) parameters - Cmax | At Cycle 1 Day 1 (C1D1) after 0 hours (each cycle is 28 days)
  Phase II PK parameter
  Cmax is maximum concentration. Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Cmax | At Cycle 1 Day 1 (C1D1) after 1 hour (each cycle is 28 days)
  Phase II PK parameter
  Cmax is maximum concentration. Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Cmax | At Cycle 1 Day 1 (C1D1) after 4 hours (each cycle is 28 days)
  Phase II PK parameter
  Cmax is maximum concentration. Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Cmax | At Cycle 1 Day 7 (C1D7) (each cycle is 28 days)
  Phase II PK parameter
  Cmax is maximum concentration. Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Cmax | At Cycle 2 Day 1 (C2D1) after 0 hours (each cycle is 28 days)
  Phase II PK parameter
  Cmax is maximum concentration. Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Cmax | At Cycle 2 Day 1 (C2D1) after 1 hour (each cycle is 28 days)
  Phase II PK parameter
  Cmax is maximum concentration. Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Cmax | At Cycle 4 Day 1 (C4D1) after 0 hours (each cycle is 28 days)
  Phase II PK parameter
  Cmax is maximum concentration. Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Cmax | At Cycle 4 Day 1 (C4D1) after 1 hour (each cycle is 28 days)
  Phase II PK parameter
  Cmax is maximum concentration. Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Ctrough | At Cycle 1 Day 1 (C1D1) after 0 hours (each cycle is 28 days)
  Phase II PK parameter
  Ctrough is lowest concertration of Inotuzumab in the blood.Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Ctrough | At Cycle1 Day 1 (C1D1) after 1 hour (each cycle is 28 days)
  Phase II PK parameter
  Ctrough is lowest concertration of Inotuzumab in the blood.Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Ctrough | At Cycle1 Day 1 (C1D1) after 4 hours (each cycle is 28 days)
  Phase II PK parameter
  Ctrough is lowest concertration of Inotuzumab in the blood.Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Ctrough | At Cycle 1 Day 7 (C1D7) (each cycle is 28 days)
  Phase II PK parameter
  Ctrough is lowest concertration of Inotuzumab in the blood.Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Ctrough | At Cycle 2 Day 1 (C2D1) after 0 hours (each cycle is 28 days)
  Phase II PK parameter
  Ctrough is lowest concertration of Inotuzumab in the blood.Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Ctrough | At Cycle 2 Day 1 (C2D1) after 1 hour (each cycle is 28 days)
  Phase II PK parameter
  Ctrough is lowest concertration of Inotuzumab in the blood.Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Ctrough | At Cycle 4 Day 1 (C4D1) after 0 hours (each cycle is 28 days)
  Phase II PK parameter
  Ctrough is lowest concertration of Inotuzumab in the blood.Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.
Phase II pharmacokinetic (PK) parameters - Ctrough | At Cycle 4 Day 1 (C4D1) after 1 hour (each cycle is 28 days)
  Phase II PK parameter
  Ctrough is lowest concertration of Inotuzumab in the blood.Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean, its associated geometric %CV) of inotuzumab ozogamicin serum concentrations will be presented in tabular form by cycle, day, and nominal time for the PK concentration analysis population.

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (7):
- United States (7):
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio

REFERENCES:
- [Derived] Metheny LL, Sobecks R, Cho C, Fu P, Margevicius S, Wang J, Ciarrone L, Kopp S, Convents RD, Majhail N, Caimi PF, Otegbeye F, Cooper BW, Gallogly M, Malek E, Tomlinson B, Gerds AT, Hamilton B, Giralt S, Perales MA, de Lima M. A multicenter study of posttransplantation low-dose inotuzumab ozogamicin to prevent relapse of acute lymphoblastic leukemia. Blood Adv. 2024 Mar 26;8(6):1384-1391. doi: 10.1182/bloodadvances.2023011514. PMID 38170741